CLINICAL TRIAL: NCT00635388
Title: A Double-blind, Randomized, Placebo-controlled Study of the Effects of Probiotics in Children Grades 1-3
Brief Title: A Study of the Effects of Probiotics in Children Grades 1-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Carl J Eastwood, Procter & Gamble
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2007149
Record Dates: First submitted 2008-02-19; First posted 2008-03-13 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Sham Comparator)
  Interventions: Other: Placebo
- 2 (Experimental)
  Interventions: Other: Lactobacillus (Probiotic 1)
- 3 (Experimental)
  Interventions: Other: Lactobacillus and Bifidobacterium (Probiotic 2)

INTERVENTIONS:
Other: Placebo — oral, placebo, once/day for 12 weeks
  Arms: 1
Other: Lactobacillus (Probiotic 1) — oral, Lactobacillus, once/day for 12 weeks
  Arms: 2
Other: Lactobacillus and Bifidobacterium (Probiotic 2) — oral, Lactobacillus and Bifidobacterium, once/day for 12 weeks
  Arms: 3

SUMMARY:
The primary objective of this study is to determine the appropriate study design for a full-scale claims support study to evaluate the impact of 2 probiotics on healthy days in elementary school children relative to a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health as reported by their parent(s)/legal guardian;
* Be willing to refrain from ingesting any product that contains fermented live bacteria (other than their test product) during the study as confirmed by their parent(s)/legal guardian(s);
* Be willing to continue their current dietary habits for the duration of the study as confirmed by their parent(s)/legal guardian(s)

Exclusion Criteria:

* Have a known hypersensitivity or allergy to any product ingredient to be ingested during the study, as reported by their parent(s)/legal guardian(s)

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of healthy days. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Eastwood, MS, Principal Investigator — Procter and Gamble
Locations (1):
- Research Site, Cincinnati, Ohio, United States